CLINICAL TRIAL: NCT04761263
Title: Effect of Task-oriented Circuit Training on Gait Kinematics, Pelvic Symmetry and Endurance in Children With Hemiplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Horus University (Other)
Responsible Party: Principal Investigator, Mohamed Salah El-Sayed, Principal Investigator, Horus University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: melsayed_phd2021
Record Dates: First submitted 2021-02-09; First posted 2021-02-18 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Cerebral Palsy, Spastic
Keywords: hemiplegic cerebral palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: two different groups received different interventions at the same time
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selected Physical Therapy group (Active Comparator): will receive a selected physical therapy program for 90 minutes, 3 times/week for 3 successive months.
  Interventions: Other: Selected Physical therapy program
- Task-oriented circuit training group (Experimental): Children allocated to the study group will receive the same selected physical therapy program given to the control group for 45 minutes in addition to 45 minutes task-oriented circuit training program. The frequency of the whole program will be three times per week, for three months.
  Interventions: Other: Task-oriented circuit training; Other: Selected Physical therapy program

INTERVENTIONS:
Other: Task-oriented circuit training — The task-oriented circuit training program consisted of 14 workstations. Time spent at each station will be 1.5 minutes. The children will complete the activity at one station and move to another station. The whole circuit will be completed in 21 minutes and it will be repeated twice per session with 3 minutes rest interval between the 2 circuits. Children will be encouraged to work as hard as possible at each workstation and will also be given verbal feedback and instructions aimed at improving performance. The progression of the task will be considered according to each child's ability and progressed as tolerated. Progressions include increasing the number of repetitions and increasing complexity of the exercise performed at each workstation, such as the distance reached in standing, reducing the height of the chair during sit-to stand, changing the height of blocks or by increasing speed of movement.
  Arms: Task-oriented circuit training group
Other: Selected Physical therapy program — * Facilitation of balance reactions from standing position including; standing on one leg, weight shifting from standing position, stoop and recover from standing, squat from standing and standing on balance board.
  * Facilitation of counterpoising mechanism through instructing the child to kick ball from standing position as well as catching and throwing ball with his hands.
  * Gait training activities including: walking using different obstacles (rolls, wedges, stepper) and walking up and down stairs.
  * Facilitation of protective reaction from standing position by pushing the child in different directions.
  * Facilitation of rising mechanism through changing position as well as returning back to the original position e.g.: from lying to standing and from sitting to standing.
  * Strengthening exercises for back and abdominal muscles as well as upper and lower limbs.
  * Jumping in place and jumping a board.

SUMMARY:
Statement of the problem:

Does task-oriented circuit training have an effect on kinematic parameters of gait, pelvic symmetry and trunk endurance in children with hemiplegic CP?

Purpose of the study:

This study aims to:

* Investigate the effect of exercise-based task-oriented circuit training on gait kinematics including (Stride length, step length, cadence, walking speed, ankle dorsiflexion angle in initial contact, knee extension angle in midstance and hip extension angle in terminal stance) in children with hemiplegic CP.
* Determine the effect of task-oriented circuit training on pelvic symmetry including (Anterior and lateral pelvic tilting) in children with hemiplegic CP.
* Examine the effect of task-oriented circuit training on trunk endurance including (prone plank test, timed partial curl up test, front abdominal power test and unilateral supine bridge test) in children with hemiplegic CP.

DETAILED DESCRIPTION:
Children with CP have lowered physical fitness levels because their motor impairments restrict their participation in daily physical activities. Children with hemiplegic CP may experience a variety of concomitant health conditions including, movement difficulty, postural and balance instability, muscle spasticity, difficulty with motor planning and control, and cognitive impairments. They also have diminished force generation, debilitated proprioception around the core, lack of enough harmonization in core musculature, and diminished capacity to adjust coupling between the trunk, pelvis, and hip stabilizers leading to diminished proficiency of movement.

According to the concept of motor learning, training is considered to be most effective when the training task is specific to the intended outcome, as optimal improvement in function involves the practice of task-specific activities. Due to the shift in focus on functional movements rather than muscle activity or movement patterns, there has been a task-oriented approach which is based on the system model of motor control providing motivation due to specific achievements that can be made.

Task-oriented circuit training effectively provides various sensory stimulation and promotes functional activities for stroke patients; however, more attention is becoming directed to children with CP to examine the effect of the task-oriented circuit training program on functional performance in children with CP. Therefore, the aim of this study is to determine the effect of rehabilitation delivered as a task-oriented circuit exercise program on kinematic parameters of gait, pelvic symmetry, and trunk endurance in children with hemiplegic CP.

ELIGIBILITY:
Inclusion Criteria:

* Their age will be ranged from 7-10 years.
* Their motor function will be at level I and II according to Gross Motor Function Classification System GMFCS (Palisano et al., 2008).
* The degree of spasticity will range from mild to moderate according to Modified Ashworth Scale (Bohannon and Smith, 1987).
* They will be able to follow instructions during evaluation and treatment.

Exclusion Criteria:

Children will be excluded from the study if they have:

* Other types of cerebral palsy.
* Cardiovascular or respiratory disorders.
* Botulinium muscular injection in the last 6 months
* Surgical interference in lower limbs and/or spine.
* Muscloskeletal problems or fixed deformities in the spine and/or lower extremities.
* seizures.
* Visual or hearing impairment.

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2021-02-07 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Assessing the change in Angular displacement of joints during gait cycle | at baseline and after 3 months of intervention
  assessment via using 2D gait analysis by Kinovea software in order to measure change in angular displacement of joints during gait cycle including: angle of ankle dorsiflexion at initial contact, angle of knee extension at midstance and angle of hip extension during terminal stance. All of these measurements have the same unit which is (angle in degrees)
Assessing the change in Pelvic symmetry | at baseline and after 3 months of intervention
  by using palpation meter inclinometer to measure the change in anterior and lateral pelvic tilting angles in degrees
Assessing the change in spatial parameters of gait | at baseline and after 3 months of intervention
  assessment via using 2D gait analysis by Kinovea software in order to measure change in step length and stride length in centimeters.
Assessing the change in Temporal parameters of gait | at baseline and after 3 months of intervention
  assessment via using 2D gait analysis by Kinovea software in order to measure change in cadence (number of steps/minute) and walking speed (meter/minute)

SECONDARY OUTCOMES:
Assessing the change in Trunk muscles endurance | at baseline and after 3 months of intervention
  Endurance of the trunk muscles will be evaluated using four endurance tests designed to establish the change in isometric trunk muscles endurance including; prone plank test (sec), timed partial curl up test (sec), front abdominal power test (cm) and unilateral supine bridge test (sec). For each trunk endurance measure, the examiner will instruct the child to hold the test position as long as possible prior to all testing. Each position will be tested three times and the average time will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed El-Sayed, Assistant lecturer, Principal Investigator — Horus University in Egypt
Locations (1):
- Outpatient clinic, Faculty of Physical Therapy, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El-Sayed MS, Kilany A, El Shemy SA. Efficacy of Task-Oriented Circuit Training on Gait Kinematics, Pelvic Symmetry and Trunk Endurance in Children with Hemiplegia: A Randomized Controlled Trial. J Musculoskelet Neuronal Interact. 2025 Mar 1;25(1):36-46. doi: 10.22540/JMNI-25-036. PMID 40024226